CLINICAL TRIAL: NCT06004505
Title: The Effect of Vestibular Rehabilitation on Static Posturography Results in Individuals With Unilateral Vestibular Hypofunction
Brief Title: Effect of Vestibular Rehabilitation on Static Posturography Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gelisim University (Other)
Responsible Party: Principal Investigator, Begum Sultan Akar, master, Istanbul Gelisim University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: begümmaster
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Unilateral Vestibular Dysfunction Disease
Keywords: Unilateral vestibular hypofunction; balance; static posturography; vestibular rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vestibular Rehabilitation Group (Other): Vestibular rehabilitation program; Gaze consisted of stabilization, adaptation, neck and balance exercises.
  Interventions: Other: Vestibular Rehabilitation

INTERVENTIONS:
Other: Vestibular Rehabilitation — The patients received vestibular rehabilitation treatment in 4 sessions at 15-day intervals and applied the given exercise programs as home exercise in the form of 10 repetitions, 3 times a day. The exercises were performed sitting, standing and walking, respectively. Balance exercises were developed by changing the support area, support surface and arm positions. When they come to each session, the exercise programs are according to the patient's condition; alternating standing and walking forward, backward, tandem and semitandem positions.

SUMMARY:
Thirty subjects with unilateral vestibular hypofunction diagnosed by videonystagmography (VNG) were voluntarily included in the study. In addition to Static Posturography test, head thrust test, Unterberger test, bucket test, eyes open/closed tandem stance test, eyes open/closed semitandem stance test, Romberg test, one leg standing on foam floor with eyes open/closed and before vestibular rehabilitation treatment In the initial evaluations, the Visual Analogue Scale (VAS) and the Dizziness Disability Inventory (DHI) were applied to assess the severity of standing on one leg with eyes open/closed, dynamic visual acuity, vertigo, and fatigue. As a result of the study, it was concluded that vestibular rehabilitation is beneficial in patients with unilateral vestibular hypofunction and its effectiveness can be monitored with Static Posturography.

DETAILED DESCRIPTION:
Patients were re-evaluated after 8 weeks of vestibular rehabilitation and the results were compared. The vestibular rehabilitation program was changed every two weeks. During the eight-week period, the patients performed the exercise program 3 times a day with 10 repetitions of each exercise. According to the evaluation results after the treatment, there was a statistically significant improvement in static posturography, especially in the modified-CTSIB test. There was a statistically significant improvement in dynamic visual acuity, head thrust test, bucket test, standing on one leg on firm and foam ground with eyes open/closed, tandem stance test with eyes closed, and Unterberger test. Statistically significant scores were obtained in VAS and DHI results.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with unilateral vestibular hypofunction by VNG
* Individuals aged 18-65
* Normal otomicroscopic examination

Exclusion Criteria:

* Individuals with neurological disorders
* Having physical problems that may interfere with walking
* Central finding as a result of the VNG test
* Pathology in temporal bone MRI
* Having a cognitive impairment that prevents communication
* Have a severe visual impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Static Posturography | 8 weeks
  In this study, balance assessment was performed using Otometrics ICS Balance Platform Version 7.1.331 Static Posturography device. The patients were asked to take off their shoes and stand on the pressure platform, align themselves at the zero point seen on the computer screen, and stand as still as possible with their hands at their sides. Posturography, Modified Clinical Test of Sensory Interaction Balance (mCTSIB), Limits of Stability (LOS) and Balance Training included in the device are the evaluations made in the study.

SECONDARY OUTCOMES:
Videonystagmography (VNG) | 8 weeks
  It captures eye movements related to vestibular dysfunction using a video recorder surrounding the eye. Oculomotor tests are done to determine the ability to move the eye at normal speeds. Abnormal responses indicate central dysfunction. Another component of VNG, caloric test; It is a noninvasive method that allows the evaluation of vestibular function as a result of the creation of current in the endolymph by introducing water or air in the low frequency area directly to the eardrum of both ears.
Tandem Posture Test | 8 weeks
  The patient stretched one foot directly in front of the other for 30 seconds without support and tried to maintain his position without falling. The time was kept with a stopwatch.
Semitandem Posture Test | 8 weeks
  The patient stretched one foot slightly in front of the other for 30 seconds without support and tried to maintain her/his position without falling.
Romberg Test | 8 weeks
  The patient tried to maintain her position without falling for 30 seconds with her feet together, eyes closed, arms crossed over her/his shoulder.
One Leg Standing Test | 8 weeks
  The patient was asked to raise one leg while standing. From the moment he lifted his foot, the time began to be kept. The time was kept for 30 seconds. The time was stopped when the patient lowered their foot before 30 seconds. It was applied to both feet with the eye open and closed. Then it was applied on soft ground with eyes open and closed.
Head Thrust Test | 8 weeks
  This test is a simple bedside test aimed at determining the presence of unilateral canal paresis. It is performed by the examiner grasping the patient's head and turning his head to the right and left in a short, small amplitude, high acceleration. Before the movement, the patient is asked to look fixedly at the examiner's nose. If the vestibular system is intact on both sides, the patient's eyes should be facing the target when head thrust is stopped. If there is a decrease in vestibular function during rapid movements, the corrective saccade movement occurs in the eye and the head thrust test is positive.
Unterberger Test | 8 weeks
  It is an eyes-closed step test for the diagnosis of unilateral vestibular dysfunction. In this study, patients were first asked to count 10 steps with their eyes open to get used to it. Then, he was asked to count 50 steps in place with his hands at his sides and his eyes closed. If the patient turned more than 45 degrees to the right or left, the test was positive (abnormal), and straight progression without turning was considered normal.
Dynamic Visual Acuity Test | 8 weeks
  In this study, the patient was seated in a chair 3 m away from the Snellen visual chart consisting of 10 lines of letters hanging on the wall. First, the patient was asked where he could read in the table. The letters in the table are reduced from top to bottom. The patient's head was started to be turned to the right and left 1-2 times per second. Meanwhile, the patient began to read the letters in front of him from top to bottom. When he told us the line where the clarity deteriorated and he started to see blurry, the test was terminated and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru SEVER, Lecturer, Principal Investigator — Department of Physiotherapy & Rehabilitation; Gamze KILIÇ, PHD, Principal Investigator — Department of Physiotherapy & Rehabilitation; Kaan Can UYANIK, Lecturer, Principal Investigator — Department of Health Management; Cengiz ÇELİKYURT, Assistant Professor/MD, Study Director — Clinic of Otolaryngology
Locations (1):
- Güneşli Erdem Hospital, Istanbul, Bağcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No